CLINICAL TRIAL: NCT03317132
Title: Occupational Recovery After First Episode Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraser Health (Other)
Collaborators: Ministry of Social Development and Poverty Reduction, British Columbia (Other); Canadian Mental Health Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2014-119
Record Dates: First submitted 2015-05-22; First posted 2017-10-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-03

CONDITIONS: Psychosis
Keywords: Vocational, First-episode psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Individual Placement and Support (Experimental): One year of IPS Support
  Interventions: Behavioral: IPS
- Treatment as usual (No Intervention): Treatment as usual

INTERVENTIONS:
Behavioral: IPS — One year of IPS Support
  Arms: Individual Placement and Support

SUMMARY:
Background: To improve employment prospects for people in the chronic stages of mental illness, the gold standard is a program called Individual Placement and Support (IPS). Little research on IPS has been done with clients in the early stages of mental illness. This project aims to assess the incremental effectiveness of the IPS model of employment support over treatment-as-usual in a representative sample of early-psychosis clients . Method: One hundred consenting clients from the Fraser Health Early Psychosis Intervention (EPI) program will be recruited and randomly assigned to receive either one year of IPS support or treatment as usual (i.e., no IPS support but no constraints on the clients to seek other employment or related support themselves). Our primary hypothesis is that the early-psychosis clients receiving the IPS intervention will obtain and maintain more paid employment compared to the TAU (treatment as usual) group. Secondary hypotheses pertain to employment success as a function of both fixed and dynamic factors and assessing the cost-effectiveness of IPS.

DETAILED DESCRIPTION:
This primary objective of this project is to assess, in early psychosis clients, the IPS vocational support model that is the "gold standard" for patients with chronic illness. Specifically, the investigators aim to maximize the chances of employment after recovery from the first acute episode, and provide work experience that will help prevent development of the "chronic mental patient" role. Our primary objective is to assess the degree to which EPI clients randomized to the IPS model will procure competitive work more quickly, and work more days during one year of IPS support, compared to control group patients who continue to receive "treatment-as-usual" vocational services.

There are also several secondary objectives:

1. understand fixed and dynamic predictors of vocational success, which may help tailor the IPS model to subpopulations. Predictors that are fixed, but may help in client selection or IPS implementation, include premorbid IQ (intelligence quotient) and previous schooling or employment (respectively). More malleable predictors, where IPS might be offered in conjunction with other interventions, include various neurocognitive abilities and recreational alcohol/drug use;
2. assess changes in health service utilization and related costs as a consequence of improved occupational functioning; and
3. lay the groundwork for a later project that would assess the longer-term durability of employment and related benefits.

As part of routine clinical care, EPI staff (i.e. case manager or psychiatrist) often query readiness to return to or seek work. For this project, those staff will also query openness to employment support. If the client so wishes, the staff will describe the project, provide a blank copy of the consent form, and gain consent for the RA to contact them after 1-3 days. Since the clients are already well-engaged with our program, the investigators expect substantial success in recruitment and low attrition rates. As noted in the IPS principles, there are minimal restrictions: all clients assigned to the IPS group who interested in working will have access, regardless of job-readiness factors, substance use, symptom severity, cognitive impairments, treatment (non)adherence, or personal presentation.

The measurement strategy includes three sets of assessment interviews from both IPS and TAU clients. The Master's-level RA (research assistant), who will have clinical experience, will collect all data in the first two years. In the third year, a new RA with health economics skills will collect the utilization and social/recreational data, while an unpaid practicum student in Clinical Psychology completes the clinical interviews. Data collection will be blinded, i.e. the RA's will not know whether the client is in the IPS or vocational-service-as-usual group.

ELIGIBILITY:
Inclusion Criteria:

* be a client in the Fraser Health EPI Program,
* want to return to work,
* currently be on a stable therapeutic dose of anti-psychotic medication, and
* have mastery of the English language

Exclusion Criteria:

* No interest in seeking employment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2015-03; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Employment attainment | 1 year
  Whether employed (defined as having at least worked one day at a paid job)

SECONDARY OUTCOMES:
Self-reported Client Service Usage | 1 year
  Change in health service utilization as measured through a Client Service Receipt Inventory
Cost related to client service usage | 1 year
  A cost analysis of client service usage data (see outcome 2) will be conducted by a health economist
Number of days worked | 1 year
  Number of days in paid employment

CONTACTS AND LOCATIONS:
Overall Officials: David H Erickson, PhD, Principal Investigator — Fraser North Early Psychosis Program
Locations (1):
- Fraser Health: Royal Columbian Hospital, New Westminster, British Columbia, Canada